CLINICAL TRIAL: NCT06889376
Title: The Use of Intranasal Sedation With Midazolam to Reduce Stress, Discomfort and Procedural Pain in Preterm Newborns and Infants During Routine ROP Screening
Brief Title: Use of Intranasal Midazolam to Reduce Stress and Procedural Pain in Premature Infants During Routine ROP Examination.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Agnieszka Nowacka, Principal Investigator, Senior Assistant at Neonatology Department, Polish Mother Memorial Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 98/2024
Record Dates: First submitted 2025-02-19; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Drug Safety
Keywords: intranasal midazolam; ROP screening; Premature infants
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal midazolam and comfort care (Experimental): The newborn/infant qualified for the ROP screening will receive intranasal midazolam before the procedure using a nasal atomizer.
  The newborn/infant will also receive comfort care
  Interventions: Drug: Intranasal midazolam administration via the DART™ intranasal atomization device along with routine comfort care.
- Control group (No Intervention): Control Group (non-midazolam group)
  * No midazolam administered.
  * Routine comfort care

INTERVENTIONS:
Drug: Intranasal midazolam administration via the DART™ intranasal atomization device along with routine comfort care. — Intervention: Intranasal midazolam (0.2 mg/kg) administered 10 minutes before ROP screening via the DART™ intranasal atomization device.
  Comfort Measures:
  * 1 ml of 20% glucose solution orally with a pacifier, 5 min before screening.
  * Swaddling and placement under the radiant warmer.
  Monitoring:
  * Vital Signs (heart rate, respiratory rate, blood pressure, oxygen saturation monitoring before drug administration until 2 hours after).
  * Pain assessment (PIPP scale) conducted before, during, and 10 and 30 min post-procedure.
  * Modified N-PASS to assess the level of sedation conducted before, during, 10, 30 minutes 1 hour and 2 hours post-procedure
  Observations for signs of:
  * Respiratory Distress (apnoea, desaturation, increased work of breathing)
  * Cardiovascular Instability (Bradycardia, tachycardia, hypotension)
  * Neurological Symptoms (Lethargy, seizures, abnormal tone)
  * Gastrointestinal Issues (Feeding intolerance, NEC-like symptoms)
  Other Names: nasal midazolam
  Arms: Intranasal midazolam and comfort care

SUMMARY:
The goal of this study is to learn about the safety and effectiveness of intranasal midazolam in newborns and infants born prematurely, undergoing Retinopathy of Prematurity (ROP) screening.

The main question it aims to answer is:

• Does use of intranasal midazolam is a safe, quick, non-invasive medication, that reduces the pain, stress, discomfort, and other complications in patients undergoing ROP screening?

Researchers will compare the intervention group with a comparison group of the patients who will receive routine comfort care.

DETAILED DESCRIPTION:
The aim of this parallel, prospective, nonblinded randomised control trial is to assess the effectiveness and safety of intranasal midazolam administered before ROP screening using the DART™ intranasal atomization device in preterm newborns and infants.

Participants: Preterm newborns and infants eligible for routine ROP screening. Recruitment: Parental/legal guardian consent required before random assignment to either the study or control group.

Study Groups and Randomization:

Random Assignment: Block randomization will be used. • Sample Size: 40 newborns/infants (20 in control, 20 in study group).

Study intervention and monitoring:

• Study Group (midazolam group) Intervention: intranasal midazolam (0.2 mg/kg) administered 10 minutes before ROP screening via the DART™ intranasal atomization device.

Comfort Measures:

* 1 ml of 20% glucose solution orally with a pacifier, 5 minutes before screening.
* Swaddling and placement under the radiant warmer.

Monitoring:

* Vital signs: heart rate, respiratory rate, blood pressure, oxygen saturation recorded 10 minutes before screening until 2 hours post-examination.
* Pain assessment (PIPP scale) conducted before, during, and 10, 30 minutes 1 hour and 2 hours post-procedure.
* Modified N-PASS scale to assess the level of sedation conducted before, during, 10, 30 minutes 1 hour and 2 hours post-procedure.

Control Group (non-midazolam group)

* No midazolam administered.
* Comfort measures: 1 ml of 20% glucose solution orally with a pacifier 5 minutes before screening. Swaddling and placement under the radiant warmer.

Monitoring:

* Vital signs: heart rate, respiratory rate, blood pressure, oxygen saturation recorded 10 minutes before screening until 2 hours post-examination.
* Pain assessment (PIPP scale) conducted before, during, and 10, 30 minutes 1 hour and 2 hours post-procedure.

In both groups, observations for:

* Respiratory Distress (apnoea, desaturation, increased work of breathing)
* Cardiovascular Instability (Bradycardia, tachycardia, hypotension)
* Neurological Symptoms (Lethargy, seizures, abnormal tone)
* Gastrointestinal Issues (Feeding intolerance, NEC-like symptoms)
* Infections & Sepsis (Confirmed or suspected based on clinical signs)

Study Outcome Assessment:

Change in pain and stress symptoms during ROP screening, measured by the Premature Infant Pain Profile (PIPP).

Clinical safety of intranasal midazolam using a nasal atomizer (DART™ intranasal atomization device) in newborns/infants.

Assessment of sedation post intranasal midazolam administration.

ELIGIBILITY:
Inclusion Criteria:

* Newborns qualified for ophthalmologic screening examination to detect retinopathy of prematurity (ROP):

  a. Newborns/infants born before the 32 weeks of gestation and/or with a birth weight <1500 g.
* Obtaining informed consent from a parent/legal guardian.

Exclusion Criteria:

* Newborns/infants not qualified for screening ophthalmologic examination (ROP).
* Newborns/infants clinically unstable, with respiratory disorders/cardiovascular instability before the ophthalmologic examination.
* Newborns/infants with congenital developmental defects.
* Newborns/infants receiving analgesic/sedative medications for other reasons.

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-03-24 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-06 (Estimated)

PRIMARY OUTCOMES:
Pain assessment pre and post intranasal midazolam administration | PIPP Score Assessment Time Points: 5 minutes before drug administration, during drug administration, 10, 30 minutes 1 hour and 2 hours post-procedure
  Primary Endpoint:
  - Change in the occurrence of pain symptoms and stress associated with screening ophthalmologic examination (ROP).
  Use of Premature Infant Pain Profile (PIPP) score
  * Purpose: To evaluate pain and stress responses before, during, and after the procedure.
  * Scoring Components:
    * Heart rate changes.
    * Oxygen saturation levels.
    * Facial expressions (brow bulge, eye squeeze, nasolabial furrow).
    * Behavioural state (awake, fussy, crying).
    * Gestational age adjustment.

SECONDARY OUTCOMES:
Evaluation of clinical safety of intranasal midazolam using a nasal atomizer (DART™ intranasal atomisation device) in newborns/infants. | Neonatal Adverse Event Severity Scale (NAESS) will be reported up to 24 hours following drug administration.
  To accurately report the adverse events during intranasal midazolam administration using a nasal atomizer (DART™ intranasal atomisation device) in newborns/infants, the Neonatal Adverse Event Severity Scale (NAESS) will be used.
  This scale contains generic severity criteria that can occur in neonates, followed by a list of 35 specific medical conditions: neurological, cardiovascular, respiratory, gastrointestinal, infectious, general and any other symptoms
  Each of the criteria is divided into grading system:
  Grade 1 - Mild Grade 2 - Moderate Grade 3 - Severe Grade 4 - Life- threatening Grade 5 - Death Assessment of the severity of the adverse event is based on the observation of the changes in the following components: age appropriate behavioural changes, changes from the baseline in the vital signs, changes in the required care and monitoring. Only changes from the baseline condition will be considered as a reported adverse-events.
Sedation assessment after intranasal midazolam administration. | Modified N-PASS score used to assess level of sedation time points: 5 minutes before drug administration, during drug administration, 10, 30 minutess, 1 hour and 2 hours post - drug administration.
  To assess the sedation status after intranasal midazolam administration, Modified N-PASS: Neonatal Sedation Assessment Scale will be used.
  The assessment criteria of the scale include:
  * Crying/ Irritability
  * Behaviour State
  * Facial Expression
  * Extremities Tone
  * Vital Signs: HR, RR, BP, SaO2 Each of the criteria scores from 0 to -2, the sum provides a total score and note as a negative score (0 to -10).
  Deep sedation: -10 to -6 Light sedation: -5 to - 2 Normal: -1 to +3

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Gulczyńska, Professor, Study Chair — Polish Mother's Health Center Institute
Locations (1):
- Polish Mother's Health Center Institute Rzgowska 281/289, 93-338 Lodz, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salaets T, Lacaze-Masmonteil T, Hokuto I, Gauldin C, Taha A, Smits A, Thewissen L, Van Horebeek I, Shoraisham A, Mohammad K, Suzuki M, Komachi S, Michels K, Turner MA, Allegaert K, Lewis T. Prospective assessment of inter-rater reliability of a neonatal adverse event severity scale. Front Pharmacol. 2023 Sep 7;14:1237982. doi: 10.3389/fphar.2023.1237982. eCollection 2023. PMID 37745081
- [Background] Salaets T, Turner MA, Short M, Ward RM, Hokuto I, Ariagno RL, Klein A, Beauman S, Wade K, Thomson M, Roberts E, Harrison J, Quinn T, Baer G, Davis J, Allegaert K; International Neonatal Consortium. Development of a neonatal adverse event severity scale through a Delphi consensus approach. Arch Dis Child. 2019 Dec;104(12):1167-1173. doi: 10.1136/archdischild-2019-317399. Epub 2019 Sep 19. PMID 31537552
- [Background] Morgan ME, Kukora S, Nemshak M, Shuman CJ. Neonatal Pain, Agitation, and Sedation Scale's use, reliability, and validity: a systematic review. J Perinatol. 2020 Dec;40(12):1753-1763. doi: 10.1038/s41372-020-00840-7. Epub 2020 Oct 2. PMID 33009491
- [Background] Vinall J, Miller SP, Chau V, Brummelte S, Synnes AR, Grunau RE. Neonatal pain in relation to postnatal growth in infants born very preterm. Pain. 2012 Jul;153(7):1374-1381. doi: 10.1016/j.pain.2012.02.007. PMID 22704600
- [Background] COMMITTEE ON FETUS AND NEWBORN and SECTION ON ANESTHESIOLOGY AND PAIN MEDICINE. Prevention and Management of Procedural Pain in the Neonate: An Update. Pediatrics. 2016 Feb;137(2):e20154271. doi: 10.1542/peds.2015-4271. Epub 2016 Jan 25. PMID 26810788
- [Background] Snyers D, Tribolet S, Rigo V. Intranasal Analgosedation for Infants in the Neonatal Intensive Care Unit: A Systematic Review. Neonatology. 2022;119(3):273-284. doi: 10.1159/000521949. Epub 2022 Mar 1. PMID 35231912
- [Background] Pasero C. Pain assessment in infants and young children: Premature Infant Pain Profile. Am J Nurs. 2002 Sep;102(9):105-6. doi: 10.1097/00000446-200209000-00065. No abstract available. PMID 12394025
- [Background] Francis K. What Is Best Practice for Providing Pain Relief During Retinopathy of Prematurity Eye Examinations? Adv Neonatal Care. 2016 Jun;16(3):220-8. doi: 10.1097/ANC.0000000000000267. PMID 27195471
- [Background] Ballantyne M, Stevens B, McAllister M, Dionne K, Jack A. Validation of the premature infant pain profile in the clinical setting. Clin J Pain. 1999 Dec;15(4):297-303. doi: 10.1097/00002508-199912000-00006. PMID 10617258
- [Background] Brummelte S, Grunau RE, Chau V, Poskitt KJ, Brant R, Vinall J, Gover A, Synnes AR, Miller SP. Procedural pain and brain development in premature newborns. Ann Neurol. 2012 Mar;71(3):385-96. doi: 10.1002/ana.22267. Epub 2012 Feb 28. PMID 22374882
- [Background] Mitchell AJ, Green A, Jeffs DA, Roberson PK. Physiologic effects of retinopathy of prematurity screening examinations. Adv Neonatal Care. 2011 Aug;11(4):291-7. doi: 10.1097/ANC.0b013e318225a332. PMID 22123352
- [Background] Moral-Pumarega MT, Caserio-Carbonero S, De-La-Cruz-Bertolo J, Tejada-Palacios P, Lora-Pablos D, Pallas-Alonso CR. Pain and stress assessment after retinopathy of prematurity screening examination: indirect ophthalmoscopy versus digital retinal imaging. BMC Pediatr. 2012 Aug 28;12:132. doi: 10.1186/1471-2431-12-132. PMID 22928523
- [Background] Thirunavukarasu AJ, Hassan R, Savant SV, Hamilton DL. Analgesia for retinopathy of prematurity screening: A systematic review. Pain Pract. 2022 Sep;22(7):642-651. doi: 10.1111/papr.13138. Epub 2022 Jun 27. PMID 35703418
- [Background] Slevin M, Murphy JF, Daly L, O'Keefe M. Retinopathy of prematurity screening, stress related responses, the role of nesting. Br J Ophthalmol. 1997 Sep;81(9):762-4. doi: 10.1136/bjo.81.9.762. PMID 9422929